CLINICAL TRIAL: NCT05842629
Title: Improved Diagnosis of Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Horsens (Other); Department of Gynaecology and Obstetrics, Viborg Regional Hospital (Unknown); Department of Gynaecology and Obstetrics, Goedstrup Regional Hospital (Unknown); Department of Gynaecology and Obstetrics, Randers Regional Hospital (Unknown)
Responsible Party: Principal Investigator, Ina Marie Dueholm Hjorth, Medical Doctor, PhD-student, Aarhus University Hospital
Other Study IDs: adnexproject
Record Dates: First submitted 2023-03-08; First posted 2023-05-06 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Neoplasms; Ovarian Cancer; Ovarian Cysts; Adnexal Mass; Adnexal Lesion; Adnexal Carcinoma; Adnexal Neoplasm
MeSH Terms: conditions — Ovarian Neoplasms; Ovarian Cysts; Carcinoma, Skin Appendage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an adnexal lesion in the Central Denmark Region

SUMMARY:
After implementation of systematic image description of adnexal masses, we aim to improve and evaluate our use of available imaging methods and biomarkers for classifying adnexal masses and distinguishing between benign and malignant adnexal masses in the hands of clinicians in Central Denmark Region.

Secondarily, we want to improve our management of adnexal masses by evaluating the complications and longitudinal changes in conservatively managed adnexal masses.

Data is registered prospectively but analyzed retrospectively.

DETAILED DESCRIPTION:
Imaging methods include ultrasonography (US) by varied observers, Magnetic Resonance Imaging (MRI) and Positron Emission Tomography-Computed Tomography (PET-CT).

Imaging criteria are based on recommendations by the International Ovarian Tumor Analysis (IOTA) group. Educational efforts in IOTA terminology and systematic description at ultrasonography may support quality in the diagnostic process.

Patients will be diagnosed and treated according to national and regional guidelines by the local clinicians.

The project has been evaluated by the Ethical Committee in the Central Denmark Region prior to initiation.

The aim of the power calculation for estimation of sample size is to be able to detect a difference in sensitivity from 75% to 90% at a threshold of 200 for Risk of Malignancy Index (RMI) and 10% for Assessment of Different NEoplasia of the adneXa (ADNEX) model and two-step-strategy / The Ovarian-Adnexal Reporting and Data System (O-RADS). To detect a difference in sensitivity (90% for ADNEX and two-step-strategy vs 75% for RMI at a specificity of 80%) at least 103 cases of malignancy should be included (calculated by using paired proportions).

ELIGIBILITY:
Patients with an adnexal mass observed at ultrasonography.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen in hospitals in the Central Denmark Region during the project period.
Sampling Method: Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficiency of available imaging modalities by models and subjective evaluation for pre-operative diagnosis of adnexal masses | 6 months
  Accuracy measures for diagnosis of ovarian cancer: Sensitivity, specificity, positive and negative predictive values.
Area Under the Receiver Operating Characteristic Curve of ADNEX, O-RADS, two-step-strategy, Simple Rules and Risk of Malignancy Index. | 6 months
  Comparison of AUC's between models/strategies

SECONDARY OUTCOMES:
Longitudinal changes in adnexal masses | Up to 5 years
  Change in imaging characteristics, occurrence of malignancy
Complications in women with conservatively managed adnexal masses | Up to 5 years
  Incidence of torsion, rupture, spontaneous resolution, surgeries.
Observer variability | 6 months
  Inter- and intra observer variation

CONTACTS AND LOCATIONS:
Overall Officials: Ina Marie Dueholm Hjorth, MD, Principal Investigator — University of Aarhus; Ole Mogensen, DMSci, Study Director — University of Aarhus
Locations (1):
- Department of Gynaecology and Obstetrics, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Not currently planned.